CLINICAL TRIAL: NCT03230357
Title: Research on the Localization Accuracy of PICC Guided by EDUG in Real World
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Branden-edug
Record Dates: First submitted 2017-07-10; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Peripherally Inserted Central Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PICC guided by EDUG (Experimental): PICC(Peripherally Inserted Central Catheter)guided by ECG Doppler ultrasonic Guidance（EDUG),EDUG is a combination device which can be used for selecting the right vein and precise positioning for the catheter tip during the PICC cathetering.
  Interventions: Device: PICC guided by EDUG

INTERVENTIONS:
Device: PICC guided by EDUG — ECG Doppler ultrasound guidance technology (EDUG) is the combination of MST puncture and ECG technology through the use of ECG Doppler ultrasound machine and valve conduction PICC to conform the localization of EDUG technology by the study of real-world

SUMMARY:
This study is a multi-center clinical study, 3000 cases, 25 centers in the country involved, carry out the guidance of EDUG PICC standardized operation at the same period. Each center assists to use app to collect research data.The experimental data will be collected, processed and analyzed by the sponsor and the researchers, and the clinical effect of EDUG will be evaluated according to the results (like the rate of once in place, the number of adjustment times before X-ray, the length of time during the whole catheter placement, the ectopic incidence during PICC first implantation and so on, the special content can be seen in the next indicator section)

ELIGIBILITY:
Inclusion Criteria:

1. Patient≥18 years old
2. Follow the doctor's advice,patients who need to be placed PICC for the first time.
3. No serious cardiovascular diseases, such as atrial fibrillation,pulmonary heart disease and other P wave abnormalities, severe heart block, etc.
4. Patients who did not participate in other clinical studies；
5. Patients who volunteer to participate the clinical study, sign the informed consent and cooperate with the clinical follow-up.

Exclusion Criteria:

1. Patients who have partial deformity or scar formation
2. Patients whose puncture site were infected or damaged
3. Patients who have sclerosis or the cord like change of the vein
4. Patients have compressed vessel by tumor
5. Patients who are confirmed or suspected having infection, bacteremia, or sepsis related to the catheter
6. Patients whose size are not fit to insert the PICC
7. Patients who are confirmed or suspected sensitive to silica gel
8. Patients who have history of radiotherapy in the pre-insertion section
9. Patients who have history of venous thrombosis, trauma, or vascular surgery
10. Patients who have superior vena cava syndrome
11. Patients who were always not following up with the doctors
12. Patients who have severe peripheral edema
13. Patients who may be required a high flow of fluid infusion, hemodialysis, pacemaker, crutches or A-V fistulation

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-02-02 (Estimated); Study Completion 2018-08-02 (Estimated)

PRIMARY OUTCOMES:
the rate of once in place | From the date of admitting to hospital until completion of the trial, up to 6 months.
  judge weather the catheter tip location guided by the EDUG is accuracy by compare the results with the Xray

SECONDARY OUTCOMES:
the number of adjustment times before X-ray | From the date of admitting until discharge to hospital, up to 14 days.
  the totally number of adjustment times during the once operation guided by EDUG
the length of time during the whole catheter placement before X-ray | From the date of admitting until discharge to hospital, up to 14 days.
  the whole length of time during the once operation guided by EDUG
the number of cathetering times after X-ray | From the date of admitting until discharge to hospital, up to 14 days.
  the totally number of cathetering times during the operation guided by EDUG until the cather tip can be guided to the right location
record the adverse events | 0,24,48,72 hours and 7days after completing the whole cathetering operation; Every 7 days from completing the whole cathering operation until tube drawing whichever came first, assessed up to 1 year
  the adverse events including bleeding, infection , thrombosis and so on
Patient acceptance | From the date of admitting until discharge to hospital, up to 14 days.
  The patient who is in line with the discharge criteria and intends to enter the study shall record whether or not he has agreed to accept the operation plan and complete the operation
the convenience of the operation | From the date of admitting until discharge to hospital, up to 14 days.
  App questionnaire was used to collect the convenience and comfort of PICC operators

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital Of Shangdong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No